CLINICAL TRIAL: NCT01568437
Title: Is the Analgesic Effect of the Transversus Abdominis Plane (TAP) Block in Laparoscopic Gastric-bypass Surgery Useful?
Brief Title: Transversus Abdominis Plane (TAP) Block in Laparoscopic Gastric-bypass Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 11-0869-B
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Gastric-bypass Surgery; Opioid Consumption; Obesity
Keywords: Laparoscopic gastric-bypass surgery; TAP block
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional management (Active Comparator): On the ward, patients will be prescribed acetaminophen 1 g every 6 hours. If additional analgesia is required, patients will take oxycodone 5-10 mg up to every 2 hours or iv morphine. Patients with contraindications to oxycodone will be prescribed oral hydromorphone 1-2 mg instead. This is the current standard of care at Toronto Western Hospital.
  Interventions: Other: Conventional Managment
- TAP Block+Conventional Management (Experimental): The TAP block will be performed after the induction, before the surgery, by an anesthesiologist with experience of at least 10 successful TAP blocks.Also patients will be prescribed acetaminophen 1 g every 6 hours. If additional analgesia is required, patients will take oxycodone 5-10 mg(oral hydromorphone 1-2 mg) up to every 2 hours or iv morphine.
  Interventions: Procedure: TAP-Block

INTERVENTIONS:
Procedure: TAP-Block — Block needle will be inserted out-of-plane to the ultrasound beam, perpendicular to the skin surface, until the tip lies deep between the fascia of the transversus abdominis muscle and the internal oblique muscle. 30 ml of the study solution in each side will be injected at this location and should be observed to spread in an anterior-posterior direction between two muscles. Each patient will receive a total dose of 60 ml of 0.25% bupivacaine (150 mg) + 1:200,000 epinephrine.
  Arms: TAP Block+Conventional Management
Other: Conventional Managment — For these group.no TAP block administration. just conventional management for post operative pain.
  Arms: Conventional management

SUMMARY:
Laparoscopic gastric-bypass surgery (LGBS) is one of the surgical treatments for morbid obesity, which is performed under general anesthesia. TAP block is an analgesic strategy covering the dermatomes from T6 to L1 and consists of injecting local anesthetic in the TAP between the costal margin and the iliac crest, where the thoracolumbar nerves (T6-L1) are located. As far as the investigators know, this analgesic technique has never been studied in LGBS. The investigators objective is to determine whether an ultrasound (US)-guided TAP block provides improved analgesia during the first 24 hours after laparoscopic gastric-bypass surgery, compared to conventional therapy only.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III
* 18-70 years of age, inclusive
* scheduled for elective laparoscopic gastric-bypass surgery.

Exclusion Criteria:

* contraindications to regional blockade (e.g., allergy to local anesthetics, coagulopathy, malignancy or infection in the area)
* pregnancy
* history of alcohol or drug dependence/abuse
* history of long term opioid intake or chronic pain disorder
* history of significant psychiatric conditions that may affect patient assessment
* inability to understand the informed consent and demands of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Opioid consumption over the first 24 hours following LGBS. | 24 hrs
  Opioid consumption will be expressed in terms of milligrams doses of PO morphine. If other opioids are used, doses will be converted to the equivalent PO morphine dose using standard opioid dosage conversion tables.

SECONDARY OUTCOMES:
Pain scores | 48 hours
  Measured with a visual analogue scale (VAS, from 0 to 10), in the postoperative care unit, at rest and on movement (coughing).
Opioid consumption at 48 hours | 48 Hours
  Opioid consumption expressed as milligram doses of PO morphine in the postoperative care unit and at 48 hours.If other opioids are used, doses will be converted to the equivalent PO morphine dose using standard opioid dosage conversion tables
Duration of block | 48 hours
  starting after block administration till drop in sensory block injection
Block procedure time | 30 minutes
  the time from placement of the ultrasound probe on the patient on one side to withdrawal of the needle on the other side;
TAP block complications | 48 hours
  vascular puncture, intravascular local anesthetic injection and local hematoma;
incidence of nausea and vomiting, and number of antiemetic medication administrations | during hospital stay average of 2 - 3 days
incidence of itching, and number of antipruritic medication administrations | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brull, MD, FRCPC, Principal Investigator — University of Toronto. University Health Network. Toronto Western Hospital.
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada